CLINICAL TRIAL: NCT06295926
Title: A Single-arm Phase II Clinical Trial of Serplulimab Combined With Concurrent Chemoradiotherapy for Limited-stage Small Cell Lung Cancer(LS-SCLC).
Brief Title: Serplulimab Combined With CCRT for LS-SCLC.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K5236
Record Dates: First submitted 2024-01-27; First posted 2024-03-06 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Etoposide; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Concurrent radiotherapy with chemotherapy (Etoposide+Cisplatin/Carboplatin) with Serplulimab, and followed by consolidation Serplulimab
  Interventions: Drug: Serplulimab

INTERVENTIONS:
Drug: Serplulimab — Undergo 4 cycles of synchronous radiotherapy and chemotherapy combined with Sintilimab immunotherapy, followed by Sintilimab monotherapy for maintenance treatment until disease progression or up to 1 year.
  Other Names: Concurrent radiotherapy Maintenance therapy; Etoposide; Cisplatin; Carboplatin

SUMMARY:
Small cell lung cancer(SCLC) has a poor prognosis and a relatively short overall survival time, urgently requiring innovative treatment strategies to improve the prognosis of such patients. Immunotherapy has become an important component of first-line therapy for extensive-stage small cell lung cancer (ES-SCLC). Studies have found that, compared to chemotherapy alone, the combination of Surlidumab with carboplatin and etoposide can extend the median overall survival in ES-SCLC to over 15 months. However, to date, research on the use of immunotherapy in combination with concurrent chemoradiotherapy (CCRT) in limited-stage small cell lung cancer (LS-SCLC) remains limited. This study aims to explore the clinical benefits of Surlidumab in combination with concurrent chemoradiotherapy in LS-SCLC and evaluate the safety of immunotherapy in combination with CCRT as first-line treatment for LS-SCLC. At the same time, it seeks to identify tumor-related biomarkers that can effectively predict the efficacy of immunotherapy and prognosis.

DETAILED DESCRIPTION:
The study plans to include a total of 96 patients who will receive first-line treatment consisting of 4 cycles of etoposide plus cisplatin/carboplatin and concurrent thoracic radiotherapy combined with Surlidumab immunotherapy. Following CCRT+Surlidumab treatment, patients will undergo Surlidumab consolidation therapy until disease progression or for a duration of at least 1 year. The study aims to evaluate the progression-free survival (PFS) and overall survival (OS) of patients compared to those receiving concurrent chemoradiotherapy alone, and to explore the efficacy of immunotherapy in limited-stage small cell lung cancer. Additionally, peripheral blood samples will be collected before treatment and 1 month after CCRT to explore tumor efficacy-related biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Diagnosed with small cell lung cancer by histology or cytology, and staged as limited stage (stage II-III according to the 8th edition of AJCC Cancer Staging)
3. Treatment-naïve population, not having received any prior targeted therapy, chemotherapy, radiation therapy, or immunotherapy for anti-tumor treatment
4. Measurable lesions based on RECIST 1.1
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. ECOG assessment should be conducted within 7 days prior to the first dose of the study intervention
6. Baseline hematologic, blood biochemistry, and urine biochemistry tests confirming sufficient bone marrow and organ function
7. Life expectancy of at least 6 months
8. Male participants: Male participants must agree to use effective contraception during the study treatment and for at least 180 days after the last dose, and must not donate sperm during this period
9. Female participants must not be pregnant or lactating, and must meet at least one of the following conditions:

   1. Women who are not capable of reproduction or
   2. Agree to use effective contraception during the treatment and for at least 180 days after the last dose
   3. Women capable of reproduction must undergo a serum or urine pregnancy test within 72 hours before starting the medication, and the result must be negative (minimum sensitivity 25 IU/L or equivalent units of HCG)

(11) Signed informed consent form

Exclusion Criteria:

1. Patients with extensive-stage small cell lung cancer
2. Cancer patients who have undergone surgery, radiotherapy, chemotherapy, or immunotherapy for small cell lung cancer
3. LS-SCLC patients with stage I disease amenable to surgical resection
4. Patients with active autoimmune diseases requiring systemic treatment (with disease-modifying agents, corticosteroids, or immunosuppressive drugs) within the past 2 years. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is allowed
5. History of (non-infectious) pneumonia/interstitial lung disease requiring steroids or current active pneumonia/interstitial lung disease requiring steroids
6. Previously diagnosed with immunodeficiency diseases such as immunoglobulin deficiency, aplastic anemia, etc.
7. Known history of human immunodeficiency virus (HIV) infection
8. Concurrent active hepatitis B (defined as HBV DNA > 500 copies) and hepatitis C virus (defined as HCV RNA (+)) infection
9. Known active tuberculosis history (tuberculin bacillus)
10. Receipt of live vaccine or attenuated live vaccine within 30 days prior to the first study intervention. Use of inactivated vaccines is allowed. Live vaccines include, but are not limited to: measles, mumps, rubella, varicella/zoster (chickenpox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccines. Injectable seasonal influenza vaccine is generally an inactivated virus vaccine and is allowed; however, intranasal influenza vaccine (e.g., FluMist®) is an attenuated live vaccine and is not allowed
11. Known other malignancy within the past 1 year that is progressing or requires active treatment. Note: Excludes adequately treated basal cell carcinoma, squamous cell skin cancer, or in situ carcinoma (excluding in situ bladder carcinoma)
12. Symptomatic central nervous system metastases and/or carcinomatous meningitis
13. Severe hypersensitivity reaction (≥3 grade) to nivolumab/platinum/etoposide and/or any of their excipients
14. Active infection requiring systemic therapy
15. Any medical condition the investigator believes would pose excessive risk to the patient. For example, poorly controlled diabetes, active infection requiring parenteral anti-infective therapy, hepatic failure, any psychiatric condition that would interfere with understanding the informed consent form (ICF). Any past or present disease, treatment, laboratory abnormality, or other condition that, in the opinion of the investigator, would confound the study results or interfere with participation throughout the study
16. Known psychiatric illness or substance abuse that would interfere with compliance with trial requirements
17. Pregnancy, lactation, planned pregnancy, or intent to become pregnant or father children during the expected duration of the study (from screening visit through 180 days after the last dose of investigational drug)
18. Prior allogeneic tissue/organ transplantation
19. Patients unable to comply with study visits
20. Currently participating in or has used other investigational drugs or devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2027-01-25 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | up to 8 weeks
  the time length from enrollment to any of the following events: disease progression with first line therapy or death from any cause. Disease progression will be assessed according to RECIST 1.1

SECONDARY OUTCOMES:
Overall survival | up to 8 weeks
  the time length from enrollment to death from any cause.
Incidence of adverse events graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | up to 8 weeks
  Evaluate adverse events of any cause, treatment-related adverse events, immune-mediated adverse events according to NCI-CTCAE V5.0
objective response rate (ORR) | up to 8 weeks
  Proportion of patients with Complete and Partial Responses to first-line therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Mengzhao Wang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Department of Respiratory and Critical Care Medicine, Peking Union Medical College Hospital, Beijing, Beijing Municipality, China